CLINICAL TRIAL: NCT00209118
Title: Paroxetine for the Prevention of IFN-Alpha Associated Depression in Patients With Chronic Hepatitis C
Brief Title: Paroxetine for the Treatment of Interferon Related Side Effects for Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrew H Miller, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0112-1998
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C; Depression; Interferon-alpha Associated Side Effects
Keywords: Hepatitis C; Interferon-alpha associated side effects; Antidepressants; Prevention
MeSH Terms: conditions — Hepatitis C; Depression | interventions — Paroxetine

INTERVENTIONS:
Drug: paroxetine

SUMMARY:
A.OVERVIEW

This is a 26 week study examining the ability of paroxetine (Paxil) to prevent the development of depression and neurotoxicity in patients receiving either 3 million units of subcutaneous IFN(interferon-alpha-2b) 3 times/week (plus ribavirin, 1000-1200 mg/d)) or PEG (polyethylene glycol) interferon-alpha-2b (1.5 micrograms/kg one time a week) and ribavirin (800 to 1,400 mg a day) for chronic hepatitis C (CHC). The IFN plasma half life (t1/2 of 24 to 34 hours) of PEG, a CHC treatment recently approved by the FDA, is significantly prolonged allowing for once a week dosing. Studies indicate that the side effect profile of the two forms of IFN-alpha treatment are very similar. CHC patients will be screened for study eligibility, and a total of 100 CHC patients between the ages of 18 and 65 years old will be enrolled across three sites (30 at Emory site and a combination of 30 from the University of Pennsylvania, Rush-Presbyterian-Saint Lukes Medical Center in Chicago and Montefiore Medical Center in New York.) Two weeks prior to treatment with subcutaneous IFN-alpha-2b, patients who meet inclusion and exclusion criteria will be stratified on the basis of a history of major depression and then randomly assigned to paroxetine or placebo in double blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years including males, females and minorities
* serum positive for either anti-HCV antibodies or HCV-RNA positive by PCR
* compensated liver disease with the following minimum hematologic and biochemical criteria: hemoglobin 3 g/dl for males; 12 g/dl for females, white blood cell count > 3,000/mm3, neutrophil count >1,5000/mm3, platelets > 100,000/mm3, prothrombin time 2 seconds prolonged compared to control, or equivalent INR ratio, albumin stable and within normal limits, serum creatinine within normal limits, thyroid-stimulating hormone (TSH) within normal limits, direct bilirubin 0.3 mg/dl or within 20% of upper limit of normal (ULN) for local laboratory, indirect bilirubin 0.8 mg/dl or within 20% of ULN for local laboratory, fasting blood sugar 115 mg/dl or within 20% of ULN for non-diabetic patients
* serum hepatitis B surface antigen (HbsAg) negative, antinuclear antibodies (ANA) 1:320
* normal pre-therapy ocular examination if a history of diabetes or hypertension
* hemoglobin A1C <8.5% if a history of diabetes
* negative pregnancy test for women of childbearing potential, and consent to adhere to adequate contraception or monogamous relationship with a male partner who has had a vasectomy during the treatment period and for 6 months after discontinuation of therapy
* not breast feeding
* documentation and confirmation of adequate contraception in sexually active males
* free from all psychotropic medications for a minimum of 14 days prior to baseline visit (8 weeks for fluoxetine)

Exclusion Criteria:

* actively meet criteria for major depression within the past six months
* active, effective treatment of depression with an antidepressant within the past three months
* meet criteria for schizophrenia or bipolar disorder (mania) past or present
* actively meet DSM IV criteria for substance abuse/dependence within the past six months
* psychotropic medications within 14 days prior to baseline visit (8 weeks for fluoxetine)
* evidence of untreated or poorly controlled endocrine, cardiovascular, hematological, renal, or neurological disease
* evidence of decompensated liver disease (such as a history or presence of ascites, bleeding varices, spontaneous encephalopathy)
* history of CNS trauma or active seizure disorder requiring medication
* any cause for liver disease other than chronic hepatitis C, such as co-infection with hepatitis B virus and/or human immunodeficiency virus, hemochromatosis, or Wilson's disease
* prior treatment with other (other than IFN-alpha or ribavirin) immunomodulatory drugs, including corticosteroids within 6 months of entry into protocol
* clinical gout
* known hypersensitivity to alpha interferon or ribavirin
* hemoglobinopathies (e.g. thalassemia)
* a positive pregnancy test
* clinically significant retinal abnormalities
* organ transplants
* a score of <24 on the Mini Mental Status Exam (MMSE)
* prior history of severe adverse events associated with paroxetine
* any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2005-07

PRIMARY OUTCOMES:
Depressive Symptom Scores
Development of Major Depression

SECONDARY OUTCOMES:
neurotoxicity
dosage reduction
discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Miller, MD, Principal Investigator — Emory University School of Medicine, Department of Psychiatry and Behavioral Sciences

REFERENCES:
- [Derived] Raison CL, Woolwine BJ, Demetrashvili MF, Borisov AS, Weinreib R, Staab JP, Zajecka JM, Bruno CJ, Henderson MA, Reinus JF, Evans DL, Asnis GM, Miller AH. Paroxetine for prevention of depressive symptoms induced by interferon-alpha and ribavirin for hepatitis C. Aliment Pharmacol Ther. 2007 May 15;25(10):1163-74. doi: 10.1111/j.1365-2036.2007.03316.x. PMID 17451562